CLINICAL TRIAL: NCT00413829
Title: Open-label, Phase II Study Assessing Immediate Effects of Lucentis®(Ranibizumab) Administered in Conjunction With Photodynamic Therapy With Visudyne® in Patients With Choroidal Neovascularization Secondary to AMD
Brief Title: Immediate Effects of Lucentis® in Conjunction With Photodynamic Therapy With Visudyne® in Exudative AMD(IECOMB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Novartis (Industry)
Responsible Party: S. Wolf, University Hospital Inselspital, Berne
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aug1202
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Age Related Macular Degeneration
Keywords: age related macular degeneration; anti-VEGF therapy
MeSH Terms: conditions — Macular Degeneration | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Intravitreal ranibizumab with photodynamic therapy

INTERVENTIONS:
Drug: Intravitreal ranibizumab with photodynamic therapy — Intravitreal injection, photodynamic therapy

SUMMARY:
This study is an evaluation of the short term effects on CNV perfusion of a same-day administration of photodynamic therapy (PDT) with Visudyne® and an intravitreal injection of Lucentis® (ranibizumab, 0.3 mg). An evaluation of the short term effects on CNV perfusion of this combined treatment is needed for better understanding of treatment effects.

DETAILED DESCRIPTION:
The primary objective is to quantify the short term effects on CNV perfusion of the same-day administration of photodynamic therapy with Visudyne® and an intravitreal injection of ranibizumab. These short term effects will be assessed with visual acuity measurements and ophthalmic examinations including indocyanine green (ICG) and fluorescein angiography (FA) as well as Optical Coherence Tomography (OCT) measurements. The primary variable for this assessment is the incidence of CNV closure one week after combined therapy as assessed with high speed ICG angiography. Fluorescein and ICG angiography will be performed using a scanning laser ophthalmoscope (HRA). All angiographic studies and OCT examinations will be evaluated by the Bern Photographic Reading Center in a masked fashion. Visual acuity assessments will be performed with Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts.

A secondary objective is to explore the effect of the same-day administration of photodynamic therapy with Visudyne® and an intravitreal injection of ranibizumab:

* on retinal thickness as measured by OCT over time
* in change of total lesion area, area of CNV assessed by FA
* in mean change of VA from baseline over time

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years of age or greater
* Patients with subfoveal choroidal neovascularization lesions secondary to AMD, either predominantly classic, occult, or minimally classic.
* CNV lesion in the study eye is ≤5400 microns in greatest linear dimension
* Patients who have a best corrected visual acuity (BCVA) score between 73 and 24 letters, inclusively, in the study eye using ETDRS-like grading charts (approximately 20/40 to 20/320) measured at 4 meters
* Willing to return for follow up scheduled visits for a 6 months period
* Only one eye will be assessed in the study. If both eyes are eligible, the one with the worse visual acuity will be selected for treatment and study unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for treatment and study

Exclusion Criteria:

* Patients who have a BCVA of < 33 letters (approximately 20/200) in both eyes
* Prior treatment in the study eye with verteporfin, external-beam radiation therapy, vitrectomy, submacular surgery, other surgical intervention for AMD, or transpupillary thermotherapy
* Previous or current intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Focal laser photocoagulation (juxta-, extra- or subfoveal ) in the study eye
* Concomitant use of chronic NSAIDs or steroids (by any route) for the duration of study participation (chronic use is defined as multiple doses taken daily for three or more consecutive days at any time during the study). Note that ASA (aspirin) taken as "low dose" up to 100 mg daily (qd) for prophylaxis of myocardial infarction (MI) and/or stroke is permitted during study
* Current use or likely need for systemic medications known to be toxic to the lens, retina or optic nerve, including Deferoxamine, Chloroquine/ hydroxychloroquine (Plaquenil), Tamoxifen, Phenothiazines and Ethambutol is excluded
* History of glaucoma filtration surgery, corneal transplant surgery or extracapsular extraction of cataract with phacoemulsification within six months preceding Day One, or a history of post-operative complications within the last 12 months preceding Day One in the study eye (uveitis, cyclitis etc.)
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with topical anti-glaucomatous medication).
* Aphakia or absence of the posterior capsule in the study eye
* Previous violation of the posterior capsule in the study eye is also excluded unless it occurred as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Presence of a retinal pigment epithelial tear involving the macula in the study eye
* Angioid streaks or precursors of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Active intraocular inflammation (grade trace or above) in the study eye
* Any active infection involving an eyeball adnexa
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
incidence of CNV closure one week after combined therapy as assessed with high speed ICG angiography | 24 months

SECONDARY OUTCOMES:
retinal thickness as measured by OCT over time | 24 months
change of total lesion area, area of CNV and area of leakage over time as assessed by FA | 24 months
mean change of VA from baseline over time | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, MD PhD, Study Chair — Klinik und Poliklinik fuer Augenheilkunde, Inselspital; Ute Wolf-Schnurrbusch, MD, Principal Investigator — Klinik und Polklinik fuer Augenheilkunde, Inselspital
Locations (1):
- Klinik und Poliklinik fuer Augenheilkunde, Inselspital, Bern, Switzerland

REFERENCES:
- [Result] Wolf-Schnurrbusch UE, Brinkmann CK, Berger L, Wolf S. Effects of combination therapy with verteporfin photodynamic therapy and ranibizumab in patients with age-related macular degeneration. Acta Ophthalmol. 2011 Sep;89(6):585-90. doi: 10.1111/j.1755-3768.2009.01747.x. Epub 2009 Oct 30. PMID 19878113